CLINICAL TRIAL: NCT03241628
Title: Generation and Evaluation of Hand Therapy Devices for Epidermolysis Bullosa (GLOVE Project): Proof of Concept Study for a Dressing Glove
Brief Title: Proof of Concept Study for a Dressing Glove
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other); Cardiff University (Other); University of Surrey (Other)
Responsible Party: Sponsor
Other Study IDs: 17/LO/0420
Record Dates: First submitted 2017-07-31; First posted 2017-08-07 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Epidermolysis Bullosa Dystrophica
Keywords: Skin blisters; Finger webbing; Finger contracture; Hand contracture
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica; Blister

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dressing Glove: Fitting bespoke dressing gloves (viscose Class 1 medical device) and evaluating dressing glove performance in the management of blisters using patient recorded outcome measures. The aim is to obtain proof of concept data for the dressing glove as an acceptable alternative to patch work dressings held in place with bandages.
  The study protocol recommends a daily change of the dressing glove but the patients also contribute their preference for frequency of dressing changes.
  Interventions: Device: Dressing Glove

INTERVENTIONS:
Device: Dressing Glove — Viscose dressing glove

SUMMARY:
Epidermolysis Bullosa (EB) is a group of genetic conditions causing extensive, painful skin blisters and wounds. Four main types of EB are recognised, which all affect the hands but those patients usually requiring hand therapy interventions have Recessive Dystrophic EB (RDEB).

The proof of concept study is part of the GLOVE (Generation and evaLuation Of hand therapy deVices for Epidermolysis bullosa) project. The project aims (i) to develop two hand therapy devices; a disposable dressing glove and splint glove to manage blisters, wounds and contractures that occur on the hands of people with RDEB (ii) to design and implement the Hand Therapy Online (HTO) electronic patient record system and (iii) to determine the cost effectiveness of the devices and the HTO system.

The proof of concept study focuses on testing the clinical performance and cost effectiveness of the dressing glove when compared with conventional dressings.

Recruited GLOVE participants will be invited to participate in the 14 week study, conducted using a quasi-experimental, n-of-1 research design. Patients who have not participated in GLOVE will also be invited to join. Participants will be asked to follow their usual dressing regime for six weeks. At week 7, they will be given several pairs of dressing gloves to replace their usual dressings, or starting to wear the glove if they avoid dressings normally and familiarise themselves. If participants usually wear their gloves to maintain their web spaces, they will wear these on top of the dressing glove to help assess compatibility.

Participants will provide feedback twice a week from week 7 on the dressing glove by answering 12 questions (TELER indicators) validated in the Pilot study (REC no: 16/LO/1046) using the HTO system. Data from the HTO system will be used by the Health Economist to determine the dressing glove and HTO's cost effectiveness.

DETAILED DESCRIPTION:
Principal research question/objective How effective is the disposable dressing glove when compared with the normal dressings and bandages used by the participants with RDEB based on 12 validated patient outcomes indicators that measure observations of hand function, device use, symptoms, and problems and limitations?

Secondary research questions Is the disposable dressing glove compatible with the SkinniesTM Web Spacer glove or any other make of glove used by the participants with RDEB to maintain their web spaces? Would you like to continue wearing the dressing glove? Is there anything else you(the participants) would like to tell us about the dressing glove?

Study design and methodology Study Design The proof of concept study of the dressing glove will be conducted using a quasi-experimental, n-of-1 research design drawn from the Medical Research Council Guidance for the design of complex interventions (MRC 2008). The reason for using this research design is due to a small sample of a small population of people with Recessive Dystrophic Epidermolysis Bullosa (RDEB). In addition, hand deformities amongst people with RDEB vary from one individual to another. Treatment and care also involve more than one intervention administered concurrently, for example wounds dressings, web-spacer gloves and splints. The researchers need to study the performance of these devices individually and together in terms of their effectiveness in delaying disease progression deformities.

The n-of-1 study design will enable investigation of the dressing glove performance against pre-determined performance criteria (12 patient recorded outcome measures on the HTO system) at the individual and group level with each participant acting as their own control.

Sample Size The sample for the GLOVE project is 14 participants. To date, seven adults and six children from pre-school age to school age have been recruited to the project from the project's two NHS sites, Guy's and St Thomas' (GSTT) NHS Foundation Trust and Great Ormond Street Hospital (GOSH) NHS Foundation Trust respectively. All the GLOVE participants will be invited to participate in the proof of concept study, subject to meeting the inclusion criteria.

Method of Recruitment The EB clinical team (GSTT; GOSH) will identify potential participants who meet the inclusion criteria for the study. The KCL research team will send a letter of invitation to these participants containing age appropriate information sheets, assent and consent forms (Letter of invitation V2 10 Jan 2017). The letter also has the contact details for the King's College Research team should the participants require further information. Participants will have a minimum of a week to decide if they would like to participate in the study. They will be invited to return the reply slip to the EB clinicians who will return them to the Chief Investigator. The EB clinicians will recruit and consent those participants who have not be involved in the GLOVE project to date. Those who have will be recruited and consented by the KCL research team. Adults (18 years and over) or their carers will be asked to provide written informed consent. Children (7-17 years) will also be asked to provide written informed consent. Their parents will also be asked to provide their written consent for their child to participate. Children aged 4-6 will be invited to provide written assent, once their parents have agreed to this. The parents will also provide their written consent, as will the parents of babies and toddlers. The consent and assent forms will be returned to the Chief Investigator at King's College London and kept in a locked cupboard, separated from the data in order to maintain data anonymity.

Conduct of the Proof of Concept Study The study will take place over 14 weeks. Participants will be asked to follow their usual dressing regime for six weeks. At week 7, they will be given several pairs of dressing gloves to familiarise themselves with. At week 8, participants will replace their usual dressings and bandages with the dressing glove or start to wear the gloves if they avoid dressings normally. If participants usually wear their gloves to maintain their web spaces, they will continue to wear these on top of the dressing glove to help assess compatibility.

Method of data collection Participants will provide feedback twice a week on the dressing glove by answering 12 questions (TELER indicators) using the Hand Therapy Online system (HTO), which is an electronic patient record system (HTO indicators V2 10 Jan 2017; Patient Guide V3). The indicators and the HTO were validated in the Pilot study (REC no: 16/LO/1046).

There are three types of measurements 1) TELER indicators, (2) physical measurements (3) measures of cost. The TELER indicators are a tool to measure observations of hand function, device use, symptoms and problems/limitations. The indicators measure clinically meaningful changes comprising an improvement, deterioration or no change in hand function from one time point to another. Each indicator is on a scale of six clinical steps or 'codes'. Code 5 is best case scenario or the treatment goal and code 0 is worst case scenario (i.e. the problem to be avoided) with codes 4, 3, 2 and 1 being clinically meaningful steps towards or away from the treatment goal.

GLOVE participants recruited to the study will be trained by the KCL researchers to use HTO system to provide feedback twice a week on the dressing glove by answering the TELER indicators for the dressing glove validated in the pilot study (REC no: 16/LO/1046).

The data from the HTO system will inform the methodology for measuring the cost effectiveness of the dressing glove.

Data analysis Numerical data analysis comprises automated calculation of patient specific index numbers within the digitised system (Deficit Index, Improvement Index, Maintenance Index, and Effectiveness Index) and two group indices (Health Status Index and Health Gain Index). An analysis of the costs of standard care versus the intervention will also be performed taking into account the use of products, time taken for wound care, and impact of wound care on daily living.

Researcher bias will be minimised by their minimal direct contact with the data collection process. In addition no attempt has been made to design out any confounding variables, thereby replicating the situations in which patients are normally treated.

Report writing and dissemination The Chief Investigator will take responsibility for writing the reports during the study and disseminating the findings, positive and negative, through publications and conference presentations.

The findings from the study will enable generalisations to be made to the wider population of RDEB patients with similar disease progression hand deformities that require the constant use of wound dressing and web-spacer gloves (Research Protocol V2 10 Jan 2017.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (over the age of seventeen) with RDEB who use or have used dressings and bandages on their hands.
2. Parents/carers of adults over the age of 17 with RDEB who use or have used dressings and bandages on their hands.
3. Parents/carers of babies, children and young people (up to the age of 17) with RDEB who use or have used dressings and bandages on their hands.
4. Babies, children and young people (age 1-17 years) with RDEB who use or have used dressings and bandages on their hands.
5. Able to communicate in English, verbally and in writing
6. Able to make an informed decision to participate and to give written consent
7. Not participating in concurrent clinical studies

Exclusion Criteria:

1. Babies aged less than 1 year old
2. Not able to communicate in English, verbally and in writing
3. Not able to make an informed decision to participate and to give written consent
4. Participating in concurrent clinical studies

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with RDEB and hand deformaties
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Effectiveness of disposable dressing glove compared with normal dressings and bandages | 14 weeks
  Dressing glove performance against pre-determined performance criteria (12 patient recorded outcome measures on the HTO system) at the individual and group level with each participant acting as their own control.

SECONDARY OUTCOMES:
Compatibility with the SkinniesTM Web Spacer glove | 14 weeks
  Determination of the compatibility of disposable dressing glove with the SkinniesTM Web Spacer glove or any other make of glove used by the participants with RDEB to maintain their web spaces

OTHER OUTCOMES:
Device preference | 14 weeks
  Would they like to continue to wear the dressing glove

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Grocott, PhD, Principal Investigator — NIHR i4i
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No